CLINICAL TRIAL: NCT02729571
Title: A Randomized, Double-blind, Dose-escalation Clinical Trial of the Safety, Reactogenicity and Immunogenicity of MTBVAC Compared to BCG Vaccine SSI, in Newborns Living in a Tuberculosis Endemic Region With a Safety Arm in Adults
Brief Title: Dose-escalation Safety and Immunogenicity Study to Compare MTBVAC to BCG in Newborns With a Safety Arm in Adults
Acronym: MTBVAC-Ph1b
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biofabri, S.L (Industry)
Collaborators: South African Tuberculosis Vaccine Initiative (Other); TuBerculosis Vaccine Initiative (Other); Triclinium Clinical Trial Project Management (Pty) Ltd. (Unknown); Universidad de Zaragoza (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MTBVAC-02
Record Dates: First submitted 2016-03-15; First posted 2016-04-06 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — MTBVAC vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- MTBVAC Group 1 (Experimental): Intervention: MTBVAC live vaccine (low dose)
  Interventions: Biological: MTBVAC
- MTBVAC Group 2 (Experimental): Intervention: MTBVAC live vaccine (middle dose)
  Interventions: Biological: MTBVAC
- MTBVAC Group 3 (Experimental): Intervention: MTBVAC live vaccine (high dose)
  Interventions: Biological: MTBVAC
- BCG Control Group (Active Comparator): Intervention: commercially available BCG live vaccine
  Interventions: Biological: BCG

INTERVENTIONS:
Biological: MTBVAC — Live-attenuated tuberculosis vaccine
  Arms: MTBVAC Group 1; MTBVAC Group 2; MTBVAC Group 3
Biological: BCG — Commercially available live-attenuated tuberculosis vaccine
  Arms: BCG Control Group

SUMMARY:
Randomized, controlled, double blind clinical trial in 2 stages (adult stage, infant stage). The first stage includes 18 HIV uninfected, QFT negative, BCG vaccinated, adult participants, randomized 1:1 to receive BCG Vaccine SSI or MTBVAC at equivalent dose (5x10E05 CFU/0.1mL) (n=9 in each group). Upon favourable safety review by the DSMB for all 18 adults up to day 28 after study vaccination, the second stage will commence in thirty-six (36) HIV unexposed, BCG naïve, newborn infants, randomized 1:3 to receive BCG Vaccine SSI or MTBVAC at one of three different dose levels ( (n=9 in each group).

DETAILED DESCRIPTION:
Adult Stage:

Eighteen (18) adult participants will be recruited and randomized equally into 1 of 2 study groups (n=9 per group): MTBVAC highest dose group (approx. 5x10E05 CFU/0.1mL) or BCG SSI standard human dose (approx. 5x10E05 CFU/0.1mL).

Safety assessments will be conducted at D0, D7, D14, D28, D56, D90, and D180 post study vaccination. A diary card will be used to collect solicited local, regional, and systemic adverse event data from D0 through D14. Reactogenicity data will be collected at each study visit. Non-serious adverse events will be collected through D28. Serious adverse events will be collected during the entire study period.

Infant Stage:

Thirty-six (36) infant participants will be recruited, randomized and allocated into 4 groups of 9 participants: BCG (single dose level 2.5 x 10E05 CFU/0.05 mL); or MTBVAC at three different dose levels (lowest 2.5x10E03 CFU/0.05mL, middle 2.5x10E04 CFU/0.05mL, highest 2.5x10E05 CFU/0.05mL).

Vaccination of neonates will be staggered by cohorts on a 3 verum : 1 control basis to allow gradual evaluation of safety and reactogenicity, as follows:

Cohort 1: 9 who receive the lowest MTBVAC dose level and 3 BCG control; Cohort 2: 9 who receive the highest MTBVAC dose level and 3 BCG control; Cohort 3: 9 who receive the highest MTBVAC dose level and 3 BCG control.

All AEs and biochemical and haematological parameters (safety data) collected up until Day 28 after vaccination of the last subject of each cohort will be reviewed by DSMB to authorize progression to the next group. Safety assessments will be conducted at D0, D7, D14, D28, D70, D90, D180 and D360 post study vaccination. A diary card will be used to collect solicited local, regional, and systemic adverse event data from D0 through D14. Reactogenicity data will be collected at each study visit. Non-serious adverse events will be collected through D28. Serious adverse events will be collected during the entire study period. Unscheduled follow-up face-to-face visits will be performed as needed for safety and adverse event management.

ELIGIBILITY:
Inclusion Criteria:

Adult stage:

Inclusion criteria:

1. Male or female, age 18 to 50 years
2. Written informed consent, including permission for access to medical records and an HIV test.
3. Available for study follow up and display a willingness and capacity to comply to study procedures.
4. In good general health, as assessed by medical history and a focused physical examination.
5. HIV test (rapid test, ELISA, or PCR) negative
6. Quantiferon®-TB Gold (Cellestis) test for latent TB infection negative within 3 weeks of enrolment
7. BCG vaccination at birth as confirmed by history or the presence of a BCG scar
8. In the case of female participants, a negative urine or serum pregnancy test at enrolment, not lactating, and willingness to use an acceptable method of contraception to avoid pregnancy for the duration of the study

Infant Stage:

Inclusion Criteria:

1. Male or female neonates within 96 hours of birth.
2. Written informed parental consent, including permission to access medical records and results of antenatal HIV tests.
3. Infant participants and their caregivers available for study follow-up and display the willingness and capacity to comply with study procedures.
4. Neonates must be in good general health as assessed by antenatal history, delivery records, and focused physical examination.
5. Birth weight more than or equal to 2500 grams.
6. Apgar score at 5 minutes more than or equal to 7.
7. A maternal HIV test result (rapid test, ELISA or PCR) taken during pregnancy must be available, documented and negative.
8. Estimated gestational age more than or equal to 38 weeks

Exclusion Criteria:

Adult stage Exclusion criteria

1. A history or evidence of an acute or chronic medical or surgical condition likely to affect the safety, reactogenicity, or immunogenicity of the investigational vaccine
2. Skin condition, bruising or birth mark at the intended injection site.
3. History or evidence of previous or current active TB disease
4. History of a household contact with active TB disease who has received less than 2 months treatment

Infant Stage Exclusion criteria:

1. Infant must not have received routine BCG vaccination prior to enrolment.
2. Antenatal, intrapartum, or postnatal medical or surgical condition that may affect the safety, reactogenicity, or immunogenicity of the investigational vaccine.
3. Maternal HIV test (rapid test, ELISA or PCR) not performed antenatally, HIV test results not available, or HIV test result known positive.
4. Maternal or other household contact with newly diagnosed or incompletely treated active TB disease.

Ages: 1 Day to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2015-09; Primary Completion 2016-09 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Safety and reactogenicity in infants and adults: includes injection site and systemic and regional adverse events, solicited and unsolicited. A diary card will be for solicited local, regional, and systemic adverse event data. | Six (6) months post-study vaccination

SECONDARY OUTCOMES:
Primary immunogenicity analysis (in infants only): Measure of frequencies and co-expression patterns of CD4 and CD8 T cells expressing specific cytokines in whole blood. | Six (6) months post-study vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Michele Tameris, MD, Principal Investigator — South African Tuberculosis Vaccine Initiative
Locations (1):
- South African Tuberculosis Vaccine Initiative, Brewelskloof Hospital, Worcester, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Spertini F, Audran R, Chakour R, Karoui O, Steiner-Monard V, Thierry AC, Mayor CE, Rettby N, Jaton K, Vallotton L, Lazor-Blanchet C, Doce J, Puentes E, Marinova D, Aguilo N, Martin C. Safety of human immunisation with a live-attenuated Mycobacterium tuberculosis vaccine: a randomised, double-blind, controlled phase I trial. Lancet Respir Med. 2015 Dec;3(12):953-62. doi: 10.1016/S2213-2600(15)00435-X. Epub 2015 Nov 17. PMID 26598141
- [Background] Aguilo N, Uranga S, Marinova D, Monzon M, Badiola J, Martin C. MTBVAC vaccine is safe, immunogenic and confers protective efficacy against Mycobacterium tuberculosis in newborn mice. Tuberculosis (Edinb). 2016 Jan;96:71-4. doi: 10.1016/j.tube.2015.10.010. Epub 2015 Nov 30. PMID 26786657
- [Background] Arbues A, Aguilo JI, Gonzalo-Asensio J, Marinova D, Uranga S, Puentes E, Fernandez C, Parra A, Cardona PJ, Vilaplana C, Ausina V, Williams A, Clark S, Malaga W, Guilhot C, Gicquel B, Martin C. Construction, characterization and preclinical evaluation of MTBVAC, the first live-attenuated M. tuberculosis-based vaccine to enter clinical trials. Vaccine. 2013 Oct 1;31(42):4867-73. doi: 10.1016/j.vaccine.2013.07.051. Epub 2013 Aug 17. PMID 23965219
- [Derived] Tameris M, Mearns H, Penn-Nicholson A, Gregg Y, Bilek N, Mabwe S, Geldenhuys H, Shenje J, Luabeya AKK, Murillo I, Doce J, Aguilo N, Marinova D, Puentes E, Rodriguez E, Gonzalo-Asensio J, Fritzell B, Thole J, Martin C, Scriba TJ, Hatherill M; MTBVAC Clinical Trial Team. Live-attenuated Mycobacterium tuberculosis vaccine MTBVAC versus BCG in adults and neonates: a randomised controlled, double-blind dose-escalation trial. Lancet Respir Med. 2019 Sep;7(9):757-770. doi: 10.1016/S2213-2600(19)30251-6. Epub 2019 Aug 12. PMID 31416768